CLINICAL TRIAL: NCT03735875
Title: A Phase Ib/II Study of Venetoclax in Combination With Quizartinib in FLT3-Mutated Acute Myelogenous Leukemia (AML)
Brief Title: Venetoclax and Quizartinib in Treating Patients With FLT3-mutated Recurrent or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to other competing trials, therefore did not go on to the Phase II portion of the study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0608; NCI-2018-02396 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0608 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-11-02; First posted 2018-11-08 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation; Recurrent Acute Myeloid Leukemia; Refractory Acute Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I: Treatment (venetoclax, quizartinib) (Experimental): Dose finding: Patients receive quizartinib PO QD on days 1-28 and venetoclax PO QD beginning on day 8 of cycle 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment beyond 24 cycles at the discretion of the treating physician.
  Interventions: Drug: Quizartinib; Drug: Venetoclax
- Phase II: Treatment (venetoclax, quizartinib) (Experimental): Patients will be treated at the established dose from the phase I portion of the study.
  Patients receive quizartinib PO QD on days 1-28 and venetoclax PO QD beginning on day 8 of cycle 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment beyond 24 cycles at the discretion of the treating physician.
  Interventions: Drug: Quizartinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Quizartinib — Given PO
  Other Names: AC-220; AC010220; AC220
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of venetoclax in combination with quizartinib and how well they work in treating patients with acute myeloid leukemia that has come back or does not respond to treatment, and who are FLT3-mutation positive. Venetoclax and quizartinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of the combination of venetoclax with quizartinib in FLT3-internal tandem duplication (ITD) mutated patients with relapsed/refractory acute myeloid leukemia (AML). (Phase Ib) II. To determine the composite complete remission (CR) (CRc) rate including CR + CRp (complete remission with incomplete platelet recovery) + CRi (complete remission with incomplete count recovery) within 3 months of treatment initiation in FLT3-ITD mutated patients with relapsed/refractory AML. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the composite CRc rate including CR + CRp + CRi within 3 months of treatment initiation in FLT3-ITD mutated patients with relapsed/ refractory AML. (Phase Ib) II. To determine the overall response rate (ORR) including CRc + partial remission (PR) within 3 months of treatment initiation in FLT3-ITD mutated patients with relapsed/refractory AML. (Phase Ib) III. To determine the duration of response (DOR), progression free survival, event-free survival (EFS), overall survival (OS), and number of patients bridged to hematopoietic stem cell transplant (HSCT) and median duration to HSCT from the initiation of the combination in FLT3-ITD mutated patients with relapsed/ refractory AML. (Phase Ib) IV. To characterize the pharmacokinetic (PK) profiles of combination therapy of venetoclax and quizartinib in FLT3-ITD mutated patients with relapsed/refractory AML. (Phase Ib) V. To determine the ORR within 3 months of treatment initiation in FLT3-ITD mutated patients with relapsed/ refractory AML. (Phase II) VI. To determine the DOR, progression-free survival (PFS), EFS, OS, and number of patients bridged to HSCT and median duration to HSCT from the initiation of the combination in FLT3-ITD mutated patients with relapsed/refractory AML. (Phase II) VII. To determine the safety and tolerability of the combination in FLT3-ITD mutated patients with relapsed/refractory AML. (Phase II)

EXPLORATORY OBJECTIVES:

I. To investigate possible relationships between baseline next generation gene sequencing and clinical response to the combination.

II. To investigate quantitative changes of FLT3-ITD allelic burden with time and the extent of pharmacodynamics biomarker (such as phosphorylated [p]-FLT3, p-ribosomal protein S6 kinase beta-1 [p70S6K], pERK, pSTAT) inhibition, and the induction of apoptosis in the bone marrow and peripheral blasts in patients treated with the combination.

III. To investigate possible relationships between baseline gene expression signatures, Bcl-2 family messenger ribonucleic acid (mRNA) and protein levels of AML blasts and/or stem cell sub-population, BH3 profiling of Bcl-2 family member dependency and ex vivo functional screen and clinical response to the combination.

IV. To analyze immune modulation including alterations in total and percent of CD3+ T-cells, total and percent of various T-cell subsets (CD4-effector, CD4-regs, CD8 cytotoxic T-cells), and total and percent of T-cell/T-cell subsets expressing specific checkpoint receptors/ligands with the combination.

V. To store and/or analyze surplus blood or tissue including bone marrow, if available, for potential future exploratory research into molecular and immune factors that may influence response to venetoclax and/or quizartinib (where response is defined broadly to include efficacy, tolerability or safety).

OUTLINE: This is a phase Ib dose-escalation study of quizartinib, followed by a phase II study.

Patients receive quizartinib orally (PO) once daily (QD) on days 1-28 and venetoclax PO QD beginning on day 8 of cycle 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment beyond 24 cycles at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 30 days and then every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* FLT3-ITD mutated patients with relapsed/refractory AML (up to four prior therapeutic regimens for AML i.e. up to salvage 4 AML), including patients who may have been previously exposed to prior FLT3-inhibitor/s other than quizartinib (stem cell transplant [SCT] or stem cell therapy for patients who previously underwent SCT/stem cell therapy in remission will not be considered a salvage regimen)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Serum direct bilirubin =< 1.5 x upper limit normal (ULN) (or =< 3.0 x ULN if deemed to be elevated due to leukemia)
* Alanine aminotransferase and/or aspartate aminotransferase (aspartate transaminase) =< 2.5 x ULN (or =< 5.0 x ULN if deemed elevated due to leukemia)
* Subjects with documented Gilbert's Syndrome may have a total bilirubin > 1.5 x ULN
* Potassium levels should be within institutional normal limits
* Magnesium levels should be within institutional normal limits
* Calcium (normalized for albumin) levels should be within institutional normal limits
* Adequate renal function as demonstrated by a serum creatinine =< 1.8
* Patients must provide written informed consent
* With the exception of patients with rapidly proliferative disease, the interval from prior treatment to time of initiation of venetoclax and quizartinib administration will be at least 14 days or at least 5 half-lives (whichever is shorter) for cytotoxic/noncytotoxic agents. The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochures, or drug-administration manuals) and will be documented in the protocol eligibility document. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions:

  * Intrathecal (IT) therapy for patients with controlled central nervous system (CNS) leukemia at the discretion of the principal investigator (PI). Controlled CNS leukemia is defined by the absence of active clinical signs of CNS disease and no evidence of CNS leukemia on the most recent 2 simultaneous cerebrospinal fluid (CSF) evaluations
  * Use of one dose of cytarabine (up to 2 g/m^2) or hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and on therapy. These medications will be recorded in the case-report form
* Baseline ejection fraction by echocardiogram (ECHO) or multigated acquisition scan (MUGA) must be >= 50%
* Women of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Women of childbearing potential must agree to have a negative serum or beta human chorionic gonadotropin (beta-hCG) pregnancy test result within 7 days prior to the first dose of study drugs and must agree to use an effective contraception method during the study and for 90 days following the last dose of the study. Men who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 90 days following the last dose of study drug

Exclusion Criteria:

* Subject has t(8;21) or inv(16) karyotype abnormalities
* Subject has acute promyelocytic leukemia (French-American-British Class M3 AML)
* Prior exposure to quizartinib at any time in the past
* Serum potassium < 3.5 mEq/L despite supplementation, or > 5.5 mEq/L. Serum magnesium above or below the institutional normal limit despite adequate management. Serum calcium (corrected for albumin levels) above or below institutional normal limit despite adequate management
* Patients with known allergy or hypersensitivity to quizartinib, venetoclax or any of their components
* Subject with a known history of being human immunodeficiency virus (HIV) positive (due to potential drug-drug interactions between antiretroviral medications and venetoclax, as well as anticipated venetoclax mechanism-based lymphopenia that may potentially increase the risk of opportunistic infections)

  * Note: HIV testing is not required
* Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or star fruit within 3 days prior to the initiation of study treatment
* Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator and/or the PI would adversely affect his/her participating in this study. Patients who have had any major surgical procedure within 14 days of day 1
* Subject has a malabsorption syndrome or other condition that precludes enteral route of administration
* Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to: a. Uncontrolled systemic infection requiring intravenous (IV) therapy (viral, bacterial or fungal). Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable. Patients with neutropenic fever considered infection related should be afebrile for at least 72 hours prior to first dose
* Subject has a history of other malignancies within 1 year prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
  * Patients on active antineoplastic or radiation therapy for a concurrent malignancy at the time of screening. Maintenance therapy, hormonal therapy, or steroid therapy for well-controlled malignancy is allowed
* Patients with a known positive hepatitis B or C infection by serology, with the exception of those with an undetectable viral load within 3 months (hepatitis B or C testing is not required prior to study entry). Subjects with serologic evidence of prior vaccination to hepatitis B virus (HBV) (i.e., hepatitis B surface antigen negative [HBs Ag-], and hepatitis B surface antibody positive [anti-HBs+]) may participate
* Female subjects who are pregnant or breastfeeding
* Impaired cardiac function including any of the following:

  * Screening electrocardiogram (ECG) with a corrected QT (QTc) > 450 msec. The QTc interval will be calculated by Fridericia's correction factor (QTcF) at screening and on day 1 prior to the first dose of quizartinib. The QTcF will be derived from the average QTcF in triplicate. If QTcF > 450 msec on day 1, quizartinib will not be given.
  * Patients with congenital long QT syndrome
  * History or presence of sustained ventricular tachycardia requiring medical intervention within 3 months prior to starting study drug
  * Any history of clinically significant ventricular fibrillation or torsades de pointes
  * Known history of second or third degree heart block (may be eligible if the patient currently has a pacemaker) within 3 months prior to starting study drug
  * Sustained heart rate of < 50/minute on screening or day 1 ECG
  * Right bundle branch block + left anterior hemiblock (i.e. bifascicular block)
  * Isolated right bundle branch block (RBBB) will not be an exclusion criterion
  * Complete left bundle branch block
  * Patients with myocardial infarction or unstable angina within 6 months prior to starting study drug
  * Congestive heart failure (CHF) New York (NY) Heart Association class III or IV within 3 months prior to starting study drug
  * Atrial fibrillation documented within 2 weeks prior to first dose of study drug
  * Patients who are actively taking CYP3A inducers. CYP3A4 inducers should be stopped at least 3 days prior to the first dose of quizartinib and are prohibited at any time on study. Moderate and strong CYP3A4 inhibitors should be stopped at least 3 days prior to the first dose of quizartinib and are prohibited during cycle 1. Moderate (but not strong) CYP3A4 inhibitors may be used with the below dose reductions of venetoclax after cycle 1. Patients may receive weak CYP3A4 inhibitors at any time on study. The venetoclax and quizartinib doses do not need to be adjusted for weak CYP3A4 inhibitors
  * Patients who require treatment with concomitant drugs that prolong QT/QTc interval. QT/QTc prolonging drugs should be stopped at least 3 days prior to the first dose of quizartinib and are prohibited at any time on study
  * Known family history of congenital long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval G Daver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants in the Phase I portion of this study were treated at dose level 0, therefore there was only one treatment arm for this study. This study did not move on to the Phase II portion of the study. Therefore, no patients were accrued on the Phase II portion of the study.
Groups:
- Phase I: Dose Level 0: Dose finding: Patients receive quizartinib PO QD on days 1-28 and venetoclax PO QD beginning on day 8 of cycle 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment beyond 24 cycles at the discretion of the treating physician.
  Quizartinib: Given PO
  Venetoclax: Given PO
- Phase II: Treatment (Venetoclax, Quizartinib): Patients will be treated at the established dose from the phase I portion of the study.
  Patients receive quizartinib PO QD on days 1-28 and venetoclax PO QD beginning on day 8 of cycle 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment beyond 24 cycles at the discretion of the treating physician.
  Quizartinib: Given PO
  Venetoclax: Given PO
Period: Overall Study
Arm/Group | Phase I: Dose Level 0 | Phase II: Treatment (Venetoclax, Quizartinib)
Started | 8 | 0
Completed | 8 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study did not move on to the Phase II portion of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level 0 | Phase II: Treatment (Venetoclax, Quizartinib) | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 5 |  | 5
  >=65 years | 3 |  | 3
Age, Continuous [Median (Full Range); unit: years] | 51 [43 to 81] |  | 51 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 4 |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 6 |  | 6
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) as Determined by Dose Limiting Toxicity (Phase Ib)
Time Frame: Up to 28 days
Population: All participants in the Phase I portion of this study were treated at dose level 0, therefore there was only one treatment arm for this study. This study did not move on to the Phase II portion of the study. Therefore, no patients were accrued on the Phase II portion of the study.
Measure: Number; unit: Milligrams (mg)
Arm/Group | Phase I: Treatment (Venetoclax, Quizartinib)
Number analyzed (Participants) | 8
Milligrams (mg) | 30

2. Secondary Outcome: Duration of Response (DOR) (Phase Ib)
Description: Response date to loss of response or last follow up.
Time Frame: Up to 4 years, 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I: Treatment (Venetoclax, Quizartinib)
Number analyzed (Participants) | 8
Months | 1.5 [0.4 to 2.3]

3. Secondary Outcome: Progression Free Survival (PFS) (Phase Ib)
Description: Time from date of treatment start until the date of progression or death from leukemia.
Time Frame: Up to 4 years, 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I: Treatment (Venetoclax, Quizartinib)
Number analyzed (Participants) | 8
Months | 2.3 [1.6 to 3.4]

4. Secondary Outcome: Event-free Survival (EFS) (Phase Ib)
Description: Time from date of treatment start until the date of failure or death from any cause.
Time Frame: Up to 4 years, 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I: Treatment (Venetoclax, Quizartinib)
Number analyzed (Participants) | 8
Months | 2.3 [1.6 to 3.4]

5. Secondary Outcome: Overall Survival (OS) (Phase Ib)
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 4 years, 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I: Treatment (Venetoclax, Quizartinib)
Number analyzed (Participants) | 8
Months | 3.7 [2.1 to 9.0]

6. Secondary Outcome: Number of Patients Bridged to Hematopoietic Stem Cell Transplant (HSCT) (Phase Ib)
Description: Participants who achieve an adequate response (OR) who proceed to receive a HSCT.
Time Frame: Up to 4 years, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Treatment (Venetoclax, Quizartinib)
Number analyzed (Participants) | 8
Participants | 0

7. Secondary Outcome: Number of Participants With a Response CR, CRp + CRi
Description: Response is defined as Complete Remission (CR), Complete Remission with Incomplete Platelet Recovery (CRp) + Complete Remission with Incomplete Hematological Recovery (CRi). CR is bone marrow regenerating normal hematopoietic cells and achieve a morphologic leukemia-free state and must have an ANC > 1 x 10^9/L and platelet count >/= 100 x 10^9/L, and normal marrow differential with < 5% blasts, and patients will be red blood cell (RBC) and platelet transfusion independent and no evidence of extramedullary leukemia. CRp is CR except for incomplete platelet recovery (< 100 × 10^9/L). CRi i sbone marrow regenerating normal hematopoietic cells with evidence of peripheral recovery with no (or only a few regenerating) circulating blasts and with a decrease of at least 50% in the percentage of blasts in the bone marrow aspirate with the total marrow blasts between 5% and 25% and meet the criteria for CR.
Time Frame: Up to 4 years, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Treatment (Venetoclax, Quizartinib)
Number analyzed (Participants) | 8
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 4 years, 6 months
Description: All participants in the Phase I portion of this study were treated at dose level 0, therefore there was only one treatment arm for this study. The study did not go on to the Phase II portion of the study. Zero participants were registered in Phase II, therefore the number of participants at risk for Serious Adverse Events, All-Cause Mortality and Other (Not Including Serious) Adverse Events is zero.
Arm/Group | Phase I: Dose Level 0 | Phase II: Treatment (Venetoclax, Quizartinib)
All-Cause Mortality (participants affected / at risk) | 2/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 7/8 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 0 (N=8) | Phase II: Treatment (Venetoclax, Quizartinib) (N=0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | NA
Lung infection (Infections and infestations) | 1 (1) | NA
Sepsis (Infections and infestations) | 1 (1) | NA
Sinusitis (Infections and infestations) | 1 (1) | NA
Pneumonia (Infections and infestations) | 1 (1) | NA
Pain (General disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 0 (N=8) | Phase II: Treatment (Venetoclax, Quizartinib) (N=0)
Abdominal pain (General disorders) | 2 (2) | NA
Alanine aminotransferase increased (Investigations) | 1 (1) | NA
Alkaline phosphatase increased (Investigations) | 1 (1) | NA
Allergic reaction (Immune system disorders) | 1 (1) | NA
Appendicitis (Infections and infestations) | 1 (1) | NA
Blood bilirubin increased (Investigations) | 1 (1) | NA
Blurred vision (Eye disorders) | 1 (1) | NA
Chills (General disorders) | 1 (1) | NA
Colitis (Gastrointestinal disorders) | 1 (1) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA
Dysphagia (Gastrointestinal disorders) | 1 (1) | NA
Ear Pain (Ear and labyrinth disorders) | 1 (1) | NA
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | NA
Esophagitis (Gastrointestinal disorders) | 1 (1) | NA
Fatigue (General disorders) | 2 (2) | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | NA
Fever (General disorders) | 2 (2) | NA
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 3 (3) | NA
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypotension (Vascular disorders) | 1 (1) | NA
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA
Paresthesia (Nervous system disorders) | 1 (1) | NA
Periorbital edema (Eye disorders) | 1 (1) | NA
Photophobia (Eye disorders) | 1 (1) | NA
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | NA
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | NA
Sepsis (Infections and infestations) | 2 (2) | NA
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | NA
Skin infection (Infections and infestations) | 2 (2) | NA
Vomiting (Gastrointestinal disorders) | 2 (2) | NA
Lung Infection (Infections and infestations) | 2 (2) | NA
Urinary Tract Infection (Infections and infestations) | 2 (2) | NA
Rash Pustular (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Facial Pain (General disorders) | 1 (1) | NA
Neck Pain (General disorders) | 1 (1) | NA
Non-Cardiac Chest Pain (General disorders) | 1 (1) | NA
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
This study was terminated early due to competing trials. All participants in the Phase I portion of this study were treated at dose level 0, therefore there was only one treatment arm for this study. This study did not move on to the Phase II portion of the study. Therefore, no patients were accrued on the Phase II portion of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03735875/Prot_SAP_000.pdf